CLINICAL TRIAL: NCT01122576
Title: A Three Arm Prospective Clinical Evaluation of Three FDA Approved Intraocular Lenses Designed to Improve Distance, Intermediate and Near Vision Following Lens Extraction.
Brief Title: Evaluation of 3 Intraocular Lenses Following Lens Extraction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 651
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Cataract
Keywords: Intra Ocular Lens; Ocular surgery; Phacoemulsification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Crystalens AO (Experimental): Eligible subjects to undergo small incision cataract surgery and were implanted with the Crystalens AO bilaterally.
  Interventions: Device: Crystalens AO
- ReSTOR (Active Comparator): Eligible subjects to undergo small incision cataract surgery and were implanted with the ReSTOR IOL bilaterally.
  Interventions: Device: ReSTOR
- Tecnis Multifocal IOL (Active Comparator): Eligible subjects to undergo small incision cataract surgery and were implanted with the Tecnis Multifocal IOL bilaterally.
  Interventions: Device: Tecnis Multifocal IOL

INTERVENTIONS:
Device: Crystalens AO — Crystalens AO surgically implanted bilaterally. Study observation up to 180 days.
  Arms: Crystalens AO
Device: ReSTOR — ReSTOR surgically implanted bilaterally. Study observation up to 180 days.
  Arms: ReSTOR
Device: Tecnis Multifocal IOL — Tecnis surgically implanted bilaterally. Study observation up to 180 days.
  Arms: Tecnis Multifocal IOL

SUMMARY:
The objective of this study is to evaluate the efficacy and subject satisfaction with three different FDA approved lenses for adults over 40 years of age who desire a reduction in spectacle dependence.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinically documented diagnosis of age-related bilateral cataracts that are considered amenable to treatment with standard phacoemulsification cataract extraction.
* Subjects must require a spherical lens power from 10.00 D to 33.00 D
* Subjects must have the potential for corrected distance visual acuity (CDVA) of 20/32 or better in both eyes, as documented by a Potential Acuity Meter

Exclusion Criteria:

* Subjects with conditions with increased risk of zonular rupture, such as pseudoexfoliation syndrome. Zonular rupture during cataract surgery may affect postoperative centration, tilt, and stability of the lens.
* Subjects who have any active inflammation or edema (swelling) of the cornea, including but not limited to the following: keratitis, keratoconjunctivitis, and keratouveitis.
* Subjects with visually significant diabetic retinopathy (proliferative or non-proliferative) which reduces potential acuity to 20/32 or worse.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omid Khodai, OD, RAC, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Inc, Aliso Viejo, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study took place at two investigative sites in the United States, with the first participant undergoing cataract surgery on 5/18/2010 and last participant completed the study on 6/27/2012.
Pre-assignment Details: Seventy eight participants (156 eyes) were enrolled in the study. 148 eyes were analyzed in both the full analysis set and the per protocol set.
Groups:
- Crystalens AO: Eligible subjects underwent small incision cataract surgery and were implanted with the Crystalens AO bilaterally.
  Crystalens AO : Crystalens AO surgically implanted bilaterally with 2 weeks between surgeries. Study observation up to 180 days.
- ReSTOR: Eligible subjects underwent small incision cataract surgery and were implanted with the ReSTOR IOL bilaterally.
  ReSTOR AOL : ReSTOR surgically implanted bilaterally with 2 weeks between surgeries. Study observation up to 180 days.
- Tecnis Multifocal IOL: Eligible subjects underwent small incision cataract surgery and were implanted with the Tecnis Multifocal IOL bilaterally.
  Tecnis Multifocal IOL :Tecnis surgically implanted bilaterally with 2 weeks between surgeries. Study observation up to 180 days.
Period: Pre-Cataract Surgery
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Started | 26 | 26 | 26
Completed | 26 | 25 | 24
Not Completed | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2
Period: Post-Cataract Surgery
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Started | 26 | 25 | 24
Completed | 26 | 25 | 22
Not Completed | 0 | 0 | 2
Not completed — Central Macular Edema | 0 | 0 | 1
Not completed — Fellow Eye Explanted | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Crystalens AO: Eligible subjects underwent small incision cataract surgery and were implanted with the Crystalens AO bilaterally.
  Crystalens AO : Crystalens AO surgically implanted bilaterally. Study observation up to 180 days.
- ReSTOR: Eligible subjects underwent small incision cataract surgery and were implanted with the ReSTOR IOL bilaterally.
  ReSTOR AOL : ReSTOR surgically implanted bilaterally. Study observation up to 180 days.
- Tecnis Multifocal IOL: Eligible subjects underwent small incision cataract surgery and were implanted with the Tecnis Multifocal IOL bilaterally.
  Tecnis Multifocal IOL : Tecnis surgically implanted bilaterally. Study observation up to 180 days.
- Total: Total of all reporting groups
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL | Total
Number analyzed (Participants) | 26 | 26 | 26 | 78
Age, Customized [Number; unit: participants]
  <40 years | 0 | 0 | 0 | 0
  40 - 49 years | 0 | 1 | 1 | 2
  50-59 years | 10 | 5 | 8 | 23
  60-69 years | 13 | 12 | 12 | 37
  70-79 years | 3 | 8 | 4 | 15
  ≥ 80 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 19 | 51
  Male | 9 | 11 | 7 | 27
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 26 | 78

OUTCOME MEASURES:

1. Primary Outcome: Mesopic Monocular Contrast Sensitivity Without Glare 1.5 and 3 Cycles/Degree
Description: Logarithm of the mesopic (low light) contrast sensitivity (ability to detect detail with subtle gradations of grayness between test target and background) without glare at five spatial frequencies (number of light and dark bars per cycle). A higher mean indicates improved contrast sensitivity
Time Frame: Postoperative visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 25 | 22
Number analyzed (eyes) | 52 | 50 | 44
log contrast sensitivity units
  1.5 cycles/degree | 1.494 (0.173) | 1.576 (0.209) | 1.410 (0.195)
  3 cycles/degree | 1.613 (0.171) | 1.679 (0.199) | 1.528 (0.175)

2. Primary Outcome: Mesopic Monocular Contrast Sensitivity Without Glare 6 Cycles/Degree
Description: as for outcome 1
Time Frame: Postoperative visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 23 | 20
Number analyzed (eyes) | 52 | 45 | 40
log contrast sensitivity units | 1.563 (0.228) | 1.644 (0.253) | 1.481 (0.212)

3. Primary Outcome: Mesopic Monocular Contrast Sensitivity Without Glare 12 Cycles/Degree
Description: as for outcome 1
Time Frame: Postoperative visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 16 | 13 | 9
Number analyzed (eyes) | 32 | 26 | 17
log contrast sensitivity units | 1.155 (0.238) | 1.335 (0.309) | 1.143 (0.189)

4. Primary Outcome: Mesopic Monocular Contrast Sensitivity Without Glare 18 Cycles/Degree
Description: as for outcome 1
Time Frame: Postoperative visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 7 | 10 | 3
Number analyzed (eyes) | 13 | 19 | 5
log contrast sensitivity units | 0.943 (0.266) | 0.950 (0.297) | 0.697 (0.138)

5. Primary Outcome: Mesopic Monocular Contrast Sensitivity Without Glare 1.5 Cycles/Degree
Description: as for outcome 1
Time Frame: Postoperative visit 4 ( 4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 25 | 22
Number analyzed (eyes) | 52 | 50 | 44
log contrast sensitivity units | 1.525 (0.203) | 1.588 (0.213) | 1.408 (0.172)

6. Primary Outcome: Mesopic Monocular Contrast Sensitivity Without Glare 3 Cycles/Degree
Description: as for outcome 1
Time Frame: Postoperative visit 4 ( 4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 25 | 22
Number analyzed (eyes) | 52 | 49 | 44
log contrast sensitivity units | 1.638 (0.243) | 1.698 (0.221) | 1.519 (0.125)

7. Primary Outcome: Mesopic Monocular Contrast Sensitivity Without Glare 6 Cycles/Degree
Description: as for outcome 1
Time Frame: Postoperative visit 4 ( 4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 25 | 24 | 21
Number analyzed (eyes) | 49 | 47 | 41
log contrast sensitivity units | 1.610 (0.241) | 1.622 (0.228) | 1.543 (0.261)

8. Primary Outcome: Mesopic Monocular Contrast Sensitivity Without Glare 12 Cycles/Degree
Description: as for outcome 1
Time Frame: Postoperative visit 4 ( 4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 17 | 15 | 8
Number analyzed (eyes) | 33 | 30 | 15
log contrast sensitivity units | 1.229 (0.262) | 1.218 (0.238) | 1.217 (0.275)

9. Primary Outcome: Mesopic Monocular Contrast Sensitivity Without Glare 18 Cycles/Degree
Description: as for outcome 1
Time Frame: Postoperative visit 4 ( 4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Groups:
- ReSTOR: Eligible subjects underwent small incision cataract surgery and wer implanted with the ReSTOR IOL bilaterally.
  ReSTOR AOL : ReSTOR surgically implanted bilaterally. Study observation up to 180 days.
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 9 | 6 | 3
Number analyzed (eyes) | 17 | 11 | 6
log contrast sensitivity units | 0.998 (0.297) | 0.789 (0.219) | 0.896 (0.275)

10. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare 1.5 & 3 Cycles/Degree
Description: as for outcome 1
Time Frame: Visit 3 (2-3 months)
Population: Full set analysis
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 25 | 25 | 20
log contrast sensitivity units
  1.5 cycles/degree | 1.688 (0.221) | 1.749 (0.201) | 1.537 (0.129)
  3 cycles/degree | 1.775 (0.252) | 1.797 (0.213) | 1.667 (0.168)

11. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare 6 Cycles/Degree
Description: as for outcome 1
Time Frame: Visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 25 | 24 | 20
log contrast sensitivity units | 1.731 (0.213) | 1.677 (0.257) | 1.593 (0.225)

12. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare 12 Cycles/Degree
Description: as for outcome 1
Time Frame: Visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 21 | 15 | 8
log contrast sensitivity units | 1.189 (0.170) | 1.362 (0.323) | 1.153 (0.228)

13. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare 18 Cycles/Degree
Description: as for outcome 1
Time Frame: Visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 7 | 10 | 3
log contrast sensitivity units | 0.965 (0.258) | 0.994 (0.359) | 0.861 (0.241)

14. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare 1.5, 3, 6 Cycles/Degree
Description: as for outcome 1
Time Frame: Visit 4 (4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 25 | 22
log contrast sensitivity units
  1.5 cycles/degree | 1.712 (0.212) | 1.743 (0.218) | 1.537 (0.147)
  3 cycles/degree | 1.785 (0.223) | 1.768 (0.243) | 1.594 (0.135)
  6 cycles/degree | 1.710 (0.234) | 1.682 (0.268) | 1.595 (0.265)

15. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare 12 Cycles/Degree
Description: as for outcome 1
Time Frame: Visit 4 (4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 18 | 17 | 9
log contrast sensitivity units | 1.261 (0.291) | 1.273 (0.269) | 1.235 (0.245)

16. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare 18 Cycles/Degree
Description: as for outcome 1
Time Frame: Visit 4 (4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 10 | 10 | 5
log contrast sensitivity units | 1.160 (0.356) | 1.008 (0.386) | 0.885 (0.287)

17. Secondary Outcome: Mesopic Monocular Contrast Sensitivity With Glare 1.5 Cycles/Degree
Description: Logarithm of the mesopic (low light) contrast sensitivity (ability to detect detail with subtle gradations of grayness between test target and background) with glare at five spatial frequencies (number of light and dark bars per cycle). A higher mean indicates improved contrast sensitivity
Time Frame: Visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 25 | 25 | 21
Number analyzed (eyes) | 50 | 49 | 42
log contrast sensitivity units | 1.329 (0.172) | 1.389 (0.219) | 1.233 (0.182)

18. Secondary Outcome: Mesopic Monocular Contrast Sensitivity With Glare 3 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 25 | 24 | 20
Number analyzed (eyes) | 50 | 48 | 39
log contrast sensitivity units | 1.527 (0.190) | 1.518 (0.267) | 1.388 (0.245)

19. Secondary Outcome: Mesopic Monocular Contrast Sensitivity With Glare 6 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 25 | 19 | 13
Number analyzed (eyes) | 49 | 38 | 27
log contrast sensitivity units | 1.514 (0.217) | 1.504 (0.313) | 1.397 (0.265)

20. Secondary Outcome: Mesopic Monocular Contrast Sensitivity With Glare 12 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 14 | 10 | 5
Number analyzed (eyes) | 27 | 20 | 10
log contrast sensitivity units | 1.118 (0.225) | 1.192 (0.235) | 1.059 (0.208)

21. Secondary Outcome: Mesopic Monocular Contrast Sensitivity With Glare 18 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 6 | 4 | 1
Number analyzed (eyes) | 11 | 8 | 1
log contrast sensitivity units | 0.883 (0.199) | 0.989 (0.336) | 0.903 (0)

22. Secondary Outcome: Mesopic Monocular Contrast Sensitivity With Glare 1.5 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 4 (4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 25 | 25 | 21
Number analyzed (eyes) | 49 | 49 | 42
log contrast sensitivity units | 1.343 (0.254) | 1.367 (0.229) | 1.199 (0.145)

23. Secondary Outcome: Mesopic Monocular Contrast Sensitivity With Glare 3 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 4 (4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 25 | 25 | 21
Number analyzed (eyes) | 49 | 49 | 41
log contrast sensitivity units | 1.536 (0.247) | 1.462 (0.212) | 1.367 (0.196)

24. Secondary Outcome: Mesopic Monocular Contrast Sensitivity With Glare 6 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 4 (4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 23 | 20 | 14
Number analyzed (eyes) | 46 | 39 | 27
log contrast sensitivity units | 1.535 (0.274) | 1.475 (0.276) | 1.413 (0.265)

25. Secondary Outcome: Mesopic Monocular Contrast Sensitivity With Glare 12 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 4 (4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 9 | 7 | 4
Number analyzed (eyes) | 18 | 14 | 7
log contrast sensitivity units | 1.341 (0.341) | 1.272 (0.358) | 1.190 (0.327)

26. Secondary Outcome: Mesopic Monocular Contrast Sensitivity With Glare 18 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 4 (4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 7 | 3 | 3
Number analyzed (eyes) | 13 | 5 | 5
log contrast sensitivity units | 1.139 (0.315) | 1.192 (0.334) | 0.849 (0.353)

27. Secondary Outcome: Mesopic Binocular Contrast Sensitivity With Glare 1.5, 3 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 24 | 25 | 19
log contrast sensitivity units
  1.5 cycles/degree | 1.459 (0.239) | 1.439 (0.216) | 1.316 (0.210)
  3 cycles/degree | 1.609 (0.189) | 1.492 (0.264) | 1.405 (0.225)

28. Secondary Outcome: Mesopic Binocular Contrast Sensitivity With Glare 6 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 24 | 20 | 15
log contrast sensitivity units | 1.574 (0.183) | 1.496 (0.385) | 1.412 (0.261)

29. Secondary Outcome: Mesopic Binocular Contrast Sensitivity With Glare 12 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 13 | 8 | 3
log contrast sensitivity units | 1.199 (0.243) | 1.337 (0.273) | 1.141 (0.222)

30. Secondary Outcome: Mesopic Binocular Contrast Sensitivity With Glare 18 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 3 (2-3 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 5 | 5 | 2
log contrast sensitivity units | 0.980 (0.295) | 1.009 (0.096) | 0.690 (0.125)

31. Secondary Outcome: Mesopic Binocular Contrast Sensitivity With Glare 1.5, 3 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 4 (4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 25 | 25 | 21
log contrast sensitivity units
  1.5 cycles/degree | 1.392 (0.222) | 1.404 (0.238) | 1.344 (0.151)
  3 cycles/degree | 1.573 (0.268) | 1.493 (0.304) | 1.410 (0.223)

32. Secondary Outcome: Mesopic Binocular Contrast Sensitivity With Glare 6 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 4 (4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 25 | 20 | 16
log contrast sensitivity units | 1.519 (0.296) | 1.515 (0.330) | 1.448 (0.271)

33. Secondary Outcome: Mesopic Binocular Contrast Sensitivity With Glare 12 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 4 (4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 9 | 8 | 2
log contrast sensitivity units | 1.321 (0.331) | 1.319 (0.450) | 1.337 (0.419)

34. Secondary Outcome: Mesopic Binocular Contrast Sensitivity With Glare 18 Cycles/Degree
Description: as for outcome 17
Time Frame: Visit 4 (4-6 months)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 6 | 5 | 2
log contrast sensitivity units | 1.175 (0.258) | 1.101 (0.439) | 1.060 (0.648)

35. Secondary Outcome: Optical Scatter
Description: Objective scatter index (OSI) was assessed using the Optical Quality Analysis System(OQAS) and summarized as a continuous variable. For this assessment, an OSI score of 1 or less represents good quality vision, 1-2 indicates some degradation but otherwise normal vision, 2-3 significant light scatter possibly requiring treatment, and scores over 4 severely compromised vision requiring intervention.
Time Frame: Visit 3 (2-3 months)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 25 | 25 | 23
Number analyzed (eyes) | 50 | 50 | 45
units on a scale | 1.1280 (0.7661) | 1.8080 (0.8685) | 1.9179 (0.9751)

36. Secondary Outcome: Optical Scatter
Description: as for outcome 35
Time Frame: Visit 4 (4-6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 25 | 22
Number analyzed (eyes) | 52 | 50 | 44
units on a scale | 1.1308 (0.7337) | 1.9760 (1.1630) | 1.8318 (0.9840)

37. Secondary Outcome: Monocular Halo and Starburst
Description: Halo and starburst (both monocular and binocular) were measured using a glarometer on integer scales of 1-5, where the smaller the number the better the outcome.
Time Frame: Visit 3 (2-3 months)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 25 | 23
Number analyzed (eyes) | 52 | 50 | 45
units on a scale
  Halo | 1.2 (0.9) | 1.3 (0.8) | 1.8 (0.9)
  Starburst | 4.5 (1.1) | 4.7 (1.0) | 4.5 (1.2)

38. Secondary Outcome: Monocular Halo and Starburst
Description: as for outcome 37
Time Frame: Visit 4 (4-6 months)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 25 | 22
Number analyzed (eyes) | 52 | 50 | 44
units on a scale
  Halo | 1.2 (0.6) | 1.5 (0.8) | 1.8 (0.7)
  Starburst | 4.6 (1.0) | 4.7 (1.0) | 4.5 (1.2)

39. Secondary Outcome: Binocular Halo and Starburst
Description: as for outcome 37
Time Frame: Visit 3 (2-3 months)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 25 | 22
units on a scale
  Halo | 1.2 (1.1) | 1.4 (0.8) | 2.0 (1.0)
  Starburst | 4.6 (1.1) | 4.7 (1.0) | 4.6 (0.9)

40. Secondary Outcome: Binocular Halo and Starburst
Description: as for outcome 37
Time Frame: Visit 4 (4-6 months)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 25 | 22
units on a scale
  Halo | 1.3 (0.7) | 1.8 (1.2) | 2.0 (0.9)
  Starburst | 4.6 (1.0) | 4.9 (0.4) | 4.5 (0.9)

41. Secondary Outcome: Manifest Refraction
Description: Manifest refraction spherical equivalent (MRSE) was calculated as the value of the sphere plus one-half of the value of the cylinder.
Time Frame: Visit 3 (2-3 Months)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 25 | 23
Number analyzed (eyes) | 52 | 50 | 45
Diopters | -0.507 (0.433) | 0.038 (0.344) | -0.114 (0.362)

42. Secondary Outcome: Manifest Refraction
Description: as for outcome 41
Time Frame: Visit 4 (4-6 Months)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 25 | 22
Number analyzed (eyes) | 52 | 50 | 44
Diopters | -0.339 (0.455) | 0.145 (0.370) | -0.091 (0.339)

43. Secondary Outcome: Uncorrected Distance Visual Acuity
Description: High Contrast Uncorrected Distance (UCDVA) measured at 32 inches, Intermediate (UCIVA) at 32 inches, and Near Visual Acuity (UCNVA) at 16 inches
Time Frame: Visit 3 (2-3 months) Visit 4 (4-6 months)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- Crystalens AO: Eligible subjects underwent small incision cataract surgery and were were implanted with the Crystalens AO bilaterally.
  Crystalens AO : Crystalens AO surgically implanted bilaterally. Study observation up to 180 days.
- ReSTOR: Eligible subjects underwent small incision cataract surgery and were were implanted with the ReSTOR IOL bilaterally.
  ReSTOR AOL : ReSTOR surgically implanted bilaterally. Study observation up to 180 days.
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 25 | 23
Number analyzed (eyes) | 52 | 50 | 46
logMAR
  UCDVA Monocular Visit 3 | 0.122 (0.171) | 0.002 (0.115) | 0.072 (0.150)
  UCDVA Monocular Visit 4 | 0.113 (0.173) | 0.016 (0.121) | 0.060 (0.148)
  UCDVA Binocular Visit 3 | 0.005 (0.082) | -0.054 (0.102) | -0.048 (0.087)
  UCDVA Binocular Visit 4 | -0.026 (0.110) | -0.061 (0.080) | -0.053 (0.104)
  UCIVA Monocular Visit 3 | 0.055 (0.159) | 0.219 (0.150) | 0.237 (0.221)
  UCIVA Monocular Visit 4 | 0.066 (0.168) | 0.244 (0.158) | 0.237 (0.197)
  UCIVA Binocular Visit 3 | -0.012 (0.130) | 0.138 (0.140) | 0.126 (0.169)
  UCIVA Binocular Visit 4 | -0.024 (0.111) | 0.169 (0.144) | 0.175 (0.146)
  UCNVA Monocular Visit 3 | 0.192 (0.189) | 0.005 (0.108) | 0.164 (0.149)
  UCNVA Monocular Visit 4 | 0.264 (0.195) | -0.008 (0.120) | 0.188 (0.185)
  UCNVA Binocular Visit 3 | 0.082 (0.151) | -0.057 (0.074) | 0.041 (0.109)
  UCNVA Binocular Visit 4 | 0.133 (0.148) | -0.061 (0.087) | 0.043 (0.130)

44. Secondary Outcome: Best-corrected Distance Visual Acuity
Description: High Contrast Distance-Corrected Distance,(BCDVA), Intermediate (DCIVA), and Near Visual Acuity (DCNVA)
Time Frame: Visit 3 (2-3 months) Visit 4 (4-6 months)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Number analyzed (Participants) | 26 | 25 | 23
Number analyzed (eyes) | 52 | 50 | 46
logMAR
  BCDVA Monocular Visit 3 | -0.100 (0.070) | -0.094 (0.080) | -0.068 (0.098)
  BCDVA Monocular Visit 4 | -0.100 (0.066) | -0.096 (0.106) | -0.075 (0.088)
  BCDVA Binocular Visit 3 | -0.144 (0.049) | -0.133 (0.073) | 0.115 (0.057)
  BCDVA Binocular Visit 4 | -0.136 (0.049) | -0.137 (0.058) | -0.117 (0.098)
  DCIVA Monocular Visit 3 | 0.169 (0.144) | 0.292 (0.132) | 0.292 (0.162)
  DCIVA Monocular Visit 4 | 0.186 (0.129) | 0.297 (0.119) | 0.328 (0.159)
  DCIVA Binocular Visit 3 | 0.095 (0.146) | 0.222 (0.112) | 0.196 (0.112)
  DCIVA Binocular Visit 4 | 0.084 (0.109) | 0.229 (0.108) | 0.229 (0.127)
  DCNVA Monocular Visit 3 | 0.346 (0.130) | -0.004 (0.087) | 0.132 (0.143)
  DCNVA Monocular Visit 4 | 0.360 (0.144) | -0.042 (0.132) | 0.136 (0.144)
  DCNVA Binocular Visit 3 | 0.261 (0.109) | -0.079 (0.065) | -0.004 (0.100)
  DCNVA Binocular Visit 4 | 0.247 (0.126) | -0.075 (0.096) | 0.025 (0.127)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Serious adverse events were measured by participant where as Other adverse events were measured by eye.
Arm/Group | Crystalens AO | ReSTOR | Tecnis Multifocal IOL
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/25 | 3/23
Other Adverse Events (participants affected / at risk) | 10/52 | 13/50 | 4/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crystalens AO (N=26) | ReSTOR (N=25) | Tecnis Multifocal IOL (N=23)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Mild vitreous hemorrhage, resolved in 38 days
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Severe central retinal vein occlusion, remained unresolved at the end of the study.
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Severe ongoing pulmonary embolism at visit 3
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — moderate pyelonephritis which was resolved in 12 days
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crystalens AO (N=52) | ReSTOR (N=50) | Tecnis Multifocal IOL (N=46)
Corneal Edema (Eye disorders) | 2 (2) | 5 (5) | 2 (2)
Punctate Keratitis (Eye disorders) | 8 (8) | 1 (1) | 2 (2)
Increased Intraocular Pressure (IOP) (Eye disorders) | 0 (0) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other